CLINICAL TRIAL: NCT05164003
Title: A Randomized, Double-blind, Active Drug Controlled, Multi-Center, Phase I/III Clinical Trial to Evaluate the Efficacy and Safety of CORETOX® in Treatment of Post Stroke Upper Limb Spasticity
Brief Title: CORETOX® in Treatment of Post Stroke Upper Limb Spasticity (Phase1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT03-KR16MST907 (Phase1)
Record Dates: First submitted 2021-12-05; First posted 2021-12-20 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity | interventions — coretox; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CORETOX® (Experimental)
  Interventions: Drug: CORETOX®
- BOTOX® (Active Comparator)
  Interventions: Drug: BOTOX®

INTERVENTIONS:
Drug: CORETOX® — Up to a total of 360U of the IP was allowed to be injected at three flexors; wrist, elbow and finger.
  Arms: CORETOX®
Drug: BOTOX® — Up to a total of 360U of the comparator was allowed to be injected at three flexors; wrist, elbow and finger.
  Arms: BOTOX®

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacodynamic of CORETOX® in the treatment of post-stroke upper limb spasticity

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 19 years

  * 6 months since the last stroke
  * 2 points in the focal spasticity of wrist flexor and ≥ 1 point at least one of elbow flexor and finger flexor as measured on MAS(0 to 4)
* Informed consent has been obtained

Exclusion Criteria:

* Neuromuscular disorders such as Lambert-Eaton syndrome, myasthenia gravis, or amyotrophic lateral sclerosis
* History(within 4 months of screening visit) or planned(during study period) treatment with phenol or alcohol injection or surgery in the target limb
* History(within 4 months of screening visit) or planned(during study period) treatment with tendon lengthening in the target limb
* Fixed joint/muscle contracture
* Severe atrophy
* Concurrent treatment with an intrathecal baclofen
* Patients who have bleeding tendency or taking anti-coagulant
* Dysphagia and Breathing Difficulties
* History(within 4 months of screening visit) Planned(during study period) treatment with Botulinum Toxin
* Known allergy or sensitivity to study medication or its components
* Concurrent or planed Muscle relaxants and/or benzodiazepine medication If patient has taken these medication stable from one month before screening and no treatment changes are not planned during the study, participation is allowed.
* Current Physical, occupational, Splinting therapy These therapy regimens will be permitted if they have been stable in the one month before screening; no treatment and no changes are planned during the study.
* Patient who are participating in other clinical trials at the screening
* Females who are pregnant, breastfeeding, or planning a pregnancy during the study period, or female of childbearing potential, not using a reliable means of contraception.
* Patients who are not eligible for this study at the discretion of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale of wrist flexor | 4 weeks
  Change from baseline at week 4 for wrist flexor muscle tone as measured on the MAS (Modified Ashworth Scale) Minimum value: 0 (best outcome) Maximum value: 4 (worst outcome)

SECONDARY OUTCOMES:
Modified Ashworth Scale of elbow and finger flexor | 4 weeks after the injection
  Change from baseline at week 4 for elbow flexor and finger flexor muscle tone as measured on MAS Minimum value: 0 (best outcome) Maximum value: 4 (worst outcome)
Modified Ashworth Scale of wrist, elbow and finger flexor | 8 and 12 weeks after the injection
  Change from baseline at week 8, 12 for wrist flexor, elbow flexor and finger flexor muscle tone as measured on MAS Minimum value: 0 (best outcome) Maximum value: 4 (worst outcome)
Modified Ashworth Scale of wrist, elbow and finger flexor | 4, 8 and 12 weeks after the injection
  The responder rate of wrist, elbow, and finger flexor tone at week 4, 8 and 12 if the responder rate is defined as at least 1-point decrease in MAS score after IP administration.
  Minimum value: 0 (best outcome) Maximum value: 4 (worst outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided